CLINICAL TRIAL: NCT06194942
Title: The EFFECT of CHIROPRACTIC THORACIC MANIPULATION on PAIN, DEPRESSION, SLEEP and QUALITY of LIFE in PATIENTS with FIBROMYALGIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, ELİF OKATAN, Physiotherapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAU-FTR-EO-01
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2023-12

CONDITIONS: Fibromyalgia
Keywords: Chiropractic, Thoracic Region, Pain, Quality of Life, Depression, Sleep
MeSH Terms: conditions — Fibromyalgia; Pain; Depression | interventions — Manipulation, Chiropractic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Other: chiropractic manipulation
- Control Group (Sham Comparator)
  Interventions: Other: sham manipulation

INTERVENTIONS:
Other: chiropractic manipulation — Chiropractic manipulation is a manual therapy technique commonly used by chiropractors. It involves the application of controlled, sudden force to a specific joint, often with the goal of improving joint function, reducing pain, and promoting overall musculoskeletal health.In the context of thoracic chiropractic manipulation, the chiropractor focuses on the vertebrae and joints in the thoracic spine.
  Arms: Treatment Group
Other: sham manipulation — Sham manipulation refers to a simulated or placebo form of a manual therapy intervention, often used in research studies, especially in clinical trials involving chiropractic or physical therapy. the term "sham manipulation" likely implies a procedure that mimics the physical aspects of a real chiropractic manipulation but does not involve the actual therapeutic forces or movements.
  The chiropractic treatment group received thoracic chiropractic manipulations (HVLA) twice a week for a total of six sessions over three weeks, while the control group received sham manipulations.
  Arms: Control Group

SUMMARY:
This study aimed to investigate the effects of thoracic chiropractic manipulations on pain intensity, depression levels, sleep, and quality of life in women diagnosed with fibromyalgia. The research included 50 female participants aged 25-45 who had been diagnosed with fibromyalgia between 2022 and 2023 at Şişli Hamidiye Etfal Education and Research Hospital. The participants were randomly divided into two groups: a chiropractic treatment group and a control group. Both groups completed pre-treatment assessments using the Visual Analog Scale (VAS), Beck Depression Inventory (BDI), Pittsburgh Sleep Quality Index (PSQI), and Short Form 36 (SF-36). The chiropractic treatment group received thoracic chiropractic manipulations (HVLA) twice a week for a total of six sessions over three weeks, while the control group received sham manipulations. A week after the final session, all participants completed the assessments again.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with fibromyalgia by a doctor.
* Having good cognitive status.
* Willingness to participate in the study voluntarily.
* Being a female aged between 25 and 45.
* The symptoms persisting without any degree of improvement or decrease recently.
* Having dysfunction (limited movement) in the thoracic region.
* Having no condition that would prevent high-velocity low-amplitude (HVLA) manipulation.

Exclusion Criteria:

* Receiving any non-pharmacological treatment.
* Having heart, kidney, or liver failure.
* Having inflammatory, psychiatric, neurological, and/or chronic progressive systemic diseases.
* Pregnancy.
* Having a history of acute or past fractures.
* Malignancy history.
* Having a history of thoracic surgery.
* Having thoracic hernias, radiculopathy, motor deficits spondylosis, spondylolisthesis, narrow canal, extruded hernia, disc herniation, discitis diagnoses.
* Metabolic bone diseases.
* Infection, fever, hypotension, respiratory disorders limiting treatment application.
* Having a rheumatic disease (except osteoarthritis).
* Osteoporosis.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
VİSUAL PAİN SCALE | before the treatment and one week after the treatment.
  he "Visual Pain Scale" is a method used to assess and quantify pain intensity through a visual representation. It typically consists of a line or numerical scale accompanied by descriptive labels or facial expressions that reflect different levels of pain severity. Participants are asked to point to or select the position on the scale that best corresponds to their perceived level of pain.

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | before the treatment and one week after the treatment.
  The Beck Depression Inventory (BDI) is a self-report questionnaire designed to assess the severity of depression symptoms in individuals.The inventory consists of 21 multiple-choice questions, each corresponding to a specific symptom of depression. Individuals are asked to select the statement that best describes their feelings over the past two weeks, including the day of the assessment. The responses are scored on a scale ranging from 0 to 3, with higher scores indicating more severe depressive symptoms. The total score can be interpreted to assess the overall level of depression, typically categorized as minimal (0-13), mild (14-19), moderate (20-28), or severe (29-63).
Pittsburgh Sleep Quality Index | before the treatment and one week after the treatment.
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire comprising 19 items, grouped into seven components, to assess various aspects of sleep quality and disturbances. Higher scores indicating poorer sleep quality.
Short Form-36 | before the treatment and one week after the treatment.
  The Short Form 36 (SF-36) is a widely used questionnaire designed to assess an individual's health-related quality of life. It consists of 36 items covering eight health domains, including physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Jülide ÖNCÜ ALPTEKİN, Professor Doctor, Study Director — Şişli Hamidiye Etfal Training and Research Hospital; Hasan Kerem ALPTEKİN, Professor Doctor, Study Director — Bahçeşehir University
Locations (1):
- Şişli Hamidiye Etfal Training and Research Hospital, Istanbul, Sarıyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Sillevis R, Cleland J, Hellman M, Beekhuizen K. Immediate effects of a thoracic spine thrust manipulation on the autonomic nervous system: a randomized clinical trial. J Man Manip Ther. 2010 Dec;18(4):181-90. doi: 10.1179/106698110X12804993427126. PMID 22131791
- [Background] Wolfe F, Walitt B, Perrot S, Rasker JJ, Hauser W. Fibromyalgia diagnosis and biased assessment: Sex, prevalence and bias. PLoS One. 2018 Sep 13;13(9):e0203755. doi: 10.1371/journal.pone.0203755. eCollection 2018. PMID 30212526
- [Background] Heidari F, Afshari M, Moosazadeh M. Prevalence of fibromyalgia in general population and patients, a systematic review and meta-analysis. Rheumatol Int. 2017 Sep;37(9):1527-1539. doi: 10.1007/s00296-017-3725-2. Epub 2017 Apr 26. PMID 28447207
- See also: Studies have demonstrated that manipulation applied to the thoracic region reduces pain and directly affects the functioning of the autonomic nervous system, given the dense connections of the autonomic nervous system in the thoracic region. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3113268/
- See also: the prevalence of Fibromyalgia Syndrome (FMS) is observed to be higher in females compared to males — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6136749/
- See also: Considering the dominance of the female gender, the study has exclusively included female patients in order to restrict gender-related factors and minimize gender-dependent influences. — https://pubmed.ncbi.nlm.nih.gov/28447207/